CLINICAL TRIAL: NCT00424632
Title: A Phase 1, Open Label, Multi-Center, Accelerated Dose-Escalation, Pharmacokinetic And Pharmacodynamic Trial Of The Oral Single Agent Aurora Kinase Inhibitor PF-03814735 In Patients With Advanced Solid Tumors For Whom No Standard Therapy Is Available
Brief Title: Phase 1 Study Of Aurora Kinase Inhibitor PF-03814735 In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9491001
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Results first posted 2012-06-12 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Solid Tumors
MeSH Terms: interventions — N-(2-(6-(4-cyclobutylamino-5-trifluoromethylpyrimidine-2-ylamino)-1,2,3,4-tetrahydro-1,4-epiazano-naphthalen-9-yl)-2-oxo-ethyl)acetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm dose escalation (Experimental)
  Interventions: Drug: PF-03814735

INTERVENTIONS:
Drug: PF-03814735 — 1, 5, and 25 mg gelatin capsules administered orally once a day from day 1 to day 5, or from day 1 to day 10 every 3 weeks until disease progression or unacceptable toxicity.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and recommended phase 2 dose of PF-03814735 administered orally as single agent in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic solid tumor resistant to standard therapy or for which no standard therapy is available
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* Brain metastases that are symptomatic and/or require treatment with steroids and/or anticonvulsants, or brain metastases that have been treated within 3 months prior to study start
* Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Nashville, Tennessee, United States
- Pfizer Investigational Site, Leuven, Belgium

REFERENCES:
- [Derived] Schoffski P, Jones SF, Dumez H, Infante JR, Van Mieghem E, Fowst C, Gerletti P, Xu H, Jakubczak JL, English PA, Pierce KJ, Burris HA. Phase I, open-label, multicentre, dose-escalation, pharmacokinetic and pharmacodynamic trial of the oral aurora kinase inhibitor PF-03814735 in advanced solid tumours. Eur J Cancer. 2011 Oct;47(15):2256-64. doi: 10.1016/j.ejca.2011.07.008. Epub 2011 Aug 16. PMID 21852114
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9491001&StudyName=Phase%201%20Study%20Of%20Aurora%20Kinase%20Inhibitor%20PF-03814735%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 59 participants enrolled and 57 sequentially assigned to treatment in Schedule A or B of study treatment. Schedule A: starting dose was 5 milligrams per day (mg/day) and dose was escalated up to 100 mg/day. Schedule B: starting dose determined based on occurrence of dose limiting toxicities and maximum tolerated dose in Schedule A.
Groups:
- PF-03814735 5 mg (Schedule A): Participants received daily dosing of PF-03814735 of 5 milligrams (mg) administered orally (PO) every morning on an empty stomach for 5 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 10 mg (Schedule A): Participants received daily dosing of PF-03814735 of 10 mg administered PO every morning on an empty stomach for 5 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 20 mg (Schedule A): Participants received daily dosing of PF-03814735 of 20 mg administered PO every morning on an empty stomach for 5 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 40 mg (Schedule A): Participants received daily dosing of PF-03814735 of 40 mg administered PO every morning on an empty stomach for 5 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 60 mg (Schedule A): Participants received daily dosing of PF-03814735 of 60 mg administered PO every morning on an empty stomach for 5 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 80 mg (Schedule A): Participants received daily dosing of PF-03814735 of 80 mg administered PO every morning on an empty stomach for 5 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 100 mg (Schedule A): Participants received daily dosing of PF-03814735 of 100 mg administered PO every morning on an empty stomach for 5 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 40 mg (Schedule B): Participants received daily dosing of PF-03814735 of 40 mg administered PO every morning on an empty stomach for 10 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 50 mg (Schedule B): Participants received daily dosing of PF-03814735 of 50 mg administered PO every morning on an empty stomach for 10 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 60 mg (Schedule B): Participants received daily dosing of PF-03814735 of 60 mg administered PO every morning on an empty stomach for 10 consecutive days out of 21-day cycles on an outpatient basis.
Period: Overall Study
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Started | 1 | 1 | 1 | 4 | 3 | 15 | 7 | 3 | 16 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 4 | 3 | 15 | 7 | 3 | 16 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Global deterioration of health status | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Objective progression or relapse | 1 | 1 | 1 | 2 | 2 | 13 | 7 | 3 | 12 | 4
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-03814735 (Schedule A): Participants received daily dosing of PF-03814735 of 5, 10, 20, 40, 60, 80, or 100 mg administered PO every morning on an empty stomach for 5 consecutive days out of 21-day cycles on an outpatient basis.
- PF-03814735 (Schedule B): Participants received daily dosing of PF-03814735 of 40, 50, or 60 mg administered PO every morning on an empty stomach for 10 consecutive days out of 21-day cycles on an outpatient basis.
- Total: Total of all reporting groups
Arm/Group | PF-03814735 (Schedule A) | PF-03814735 (Schedule B) | Total
Number analyzed (Participants) | 32 | 25 | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.0) [44 to 81] | 58.2 (10.2) [28 to 75] | 61.2 (9.8) [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Cycle Dose Limiting Toxicities (DLTs) Graded According to Common Terminology Criteria Adverse Events (CTCAE), Version 3
Description: DLT defined as any of the following during the first cycle of treatment and attributable to PF-03814735: Grade (Gr) 4 neutropenia (absolute neutrophil count [ANC] <500 cells/mm^3) for >7 days or febrile neutropenia (ANC <1000/mm^3, fever ≥38 degrees Celsius; neutropenic infection (ANC <1000/mm^3); Gr 4 thrombocytopenia (platelets <25,000 cells/mm^3); ≥Gr 3 nausea, vomiting, or diarrhea, despite optimal antiemetic, anti-diarrheal support; ≥20% decrease in left ventricular ejection fraction compared to baseline; other non-hematological toxicity; any Gr ≥3 adverse event; or failure to recover.
Time Frame: Day 1 up to Day 21 of first cycle
Population: Safety population: Same as the As-treated population, defined as all patients enrolled in the study that received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 3 | 15 | 7 | 3 | 16 | 6
participants | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: Schedule A Cycle 1/Day 4, Schedule B Cycle 1/Day 9: pre-dose, 0.5, 1, 2, 4, 6, 10, and 24 hours post-dose
Population: Pharmacokinetic (PK) parameter analysis set: Enrolled participants who received at least 1 dose of study treatment who had at least 1 of the PK parameters of interest estimated in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- PF-03814735 25 mg (Schedule B): Participant was randomized to receive daily dosing of PF-03814735 50 mg administered PO every morning on an empty stomach for 10 consecutive days out of 21-day cycles on an outpatient basis. However, participant had reduced dose of 25 mg beginning on Cycle 1 Day 1 of treatment.
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 25 mg (Schedule B) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 3 | 15 | 7 | 1 | 3 | 13 | 6
mcg/mL | 0.1920 (NA) — Geometric coefficient of variation (CV) % was not calculated for treatment groups with N <3., | 0.6470 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 0.9010 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 1.965 (35) | 3.724 (30) | 3.773 (43) | 4.106 (46) | 1.470 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 1.957 (36) | 2.786 (50) | 2.087 (24)

3. Secondary Outcome: Time for Maximum Observed Serum Concentration (Tmax)
Time Frame: Schedule A Cycle 1/Day 4, Schedule B Cycle 1/Day 9: pre-dose, 0.5, 1, 2, 4, 6, 10, and 24 hours post-dose
Population: PK parameter analysis set
Measure: Median (Full Range); unit: hours
Groups:
- PF-03814735 25 mg (Schedule B): Participant was randomized to receive daily dosing of PF-03814735 of 50 mg administered PO every morning on an empty stomach for 10 consecutive days out of 21-day cycles on an outpatient basis. However, participant had reduced dose of 25 mg beginning on Cycle 1 Day 1 of treatment.
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 25 mg (Schedule B) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 3 | 15 | 7 | 1 | 3 | 13 | 6
hours | 2.00 (NA) [2.00 to 2.00] | 1.00 (NA) [1.00 to 1.00] | 24.0 (NA) [24.0 to 24.0] | 1.50 (144) [0.500 to 6.00] | 2.00 (79) [1.00 to 4.00] | 2.00 (63) [0.500 to 4.00] | 2.00 (56) [1.00 to 4.00] | 2.00 (NA) [2.00 to 2.00] | 1.00 (79) [0.500 to 2.00] | 2.00 (59) [1.00 to 6.00] | 1.50 (61) [1.00 to 4.00]

4. Secondary Outcome: Area Under the Serum Concentration Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast)
Description: Area under the serum concentration time-curve from zero to the last measured concentration.
Time Frame: Schedule A Cycle 1/Day 4, Schedule B Cycle 1/Day 9: pre-dose, 0.5, 1, 2, 4, 6, 10, and 24 hours post-dose
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Median (Full Range); unit: mcg*hr/mL
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 25 mg (Schedule B) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Area Under the Serum Concentration Time Profile From Time 0 to Time Tau (τ), the Dosing Interval, Where τ = 24 Hours (AUCτ).
Time Frame: Schedule A Cycle 1/Day 4, Schedule B Cycle 1/Day 9: pre-dose, 0.5, 1, 2, 4, 6, 10, and 24 hours post-dose
Population: PK parameter analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 25 mg (Schedule B) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 3 | 15 | 7 | 1 | 3 | 13 | 6
mcg*hr/mL | 2.957 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 10.09 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 17.68 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 22.99 (17) | 47.95 (62) | 49.33 (58) | 57.96 (45) | 22.69 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 22.08 (90) | 37.15 (66) | 24.12 (24)

6. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin)
Description: Cmin defined as the lowest serum concentration observed during the dosing interval.
Time Frame: Schedule A Cycle 1/Day 4, Schedule B Cycle 1/Day 9: pre-dose, 0.5, 1, 2, 4, 6, 10, and 24 hours post-dose
Population: PK parameter analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 25 mg (Schedule B) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 3 | 15 | 7 | 1 | 3 | 13 | 6
mcg/mL | 0.05440 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 0.2330 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 0.3110 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 0.4521 (27) | 1.019 (105) | 1.061 (86) | 1.410 (58) | 0.4950 (NA) — Geometric CV % was not calculated for treatment groups with N <3. | 0.3901 (271) | 0.6636 (178) | 0.4217 (61)

7. Secondary Outcome: Observed Serum Accumulation Ratio (Rac)
Description: Rac was the ratio of Schedule B Cycle 1/Day 9 to Day -5 (Day 9 AUCτ to Day -5 AUCτ).
Time Frame: Schedule B Day-5: pre-dose, 0.5, 1, 2, 4, 6, 10, 24, 32, 48, and 72 hours post-dose, Schedule B Cycle 1/Day 9: pre-dose, 0.5, 1, 2, 4, 6, 10, and 24 hours post-dose
Population: PK parameter analysis set. N=number of participants in the indicated population contributing to the mean.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 3 | 13 | 6
ratio | 1.054 (28) | 1.503 (44) | 1.247 (27)

8. Secondary Outcome: Terminal Half-life (t 1/2)
Description: Terminal half-life (serum decay half-life) is the time measured for the serum concentration to decrease by one half.
Time Frame: Schedule A Cycle 1/Day 4, Schedule B Cycle 1/Day 9: pre-dose, 0.5, 1, 2, 4, 6, 10, and 24 hours post-dose
Population: Half-life (t ½) was not reported for multiple-dose data since the 24-hour sampling period was not long enough to adequately characterize t ½.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 25 mg (Schedule B) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Urine Pharmacokinetics
Description: Urine PK for quantification of unchanged PF-03814375 and any identified metabolites. 24-hour urine collection at 8-hour intervals after the morning dose (Schedule [Sch] A Day 4, Sch B Day 9; last sample collected just prior to the morning dose on Sch A Day 5 or Sch B Day 10 in the expanded maximum tolerated dose (MTD) cohort only (≥ 10 participants in Sch A 80 mg and Sch B 50 mg groups). The lower limit of quantification (LLOQ) was 1 nanogram per milliliter (ng/mL). Clinical specimens with concentrations below the LLOQ were to be reported as below the limited of quantification (BLQ) 1 ng/mL.
Time Frame: Schedule A Cycle 1/Day 4, Schedule B Cycle 1/Day 9: pre-dose, 0.5, 1, 2, 4, 6, 10, and 24 hours post-dose
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03814735 80 mg (Schedule A) | PF-03814735 50 mg (Schedule B)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Summary of Tumor Metabolism Assessed by Positron Emission Tomography With F-18-fluorodeoxyglucose (FDG-PET)
Description: FTD-PET measured as standardized uptake volume (SUV) values corrected for lean body mass. Change from baseline categorized according to European Organization for Research and Treatment for Cancer (EORTC) criteria: Partial Metabolic Response (PMR): SUV value during treatment <75 percent (%) of baseline value; Progressive Metabolic Disease (PMD): SUV value during treatment >125% of baseline value; Stable Metabolic Disease (SMD): change in SUV value between PMR and PMD. Collected in the expanded MTD cohort only (≥ 10 participants in Sch A 80 mg and Sch B 50 mg groups).
Time Frame: Baseline (Schedule A or Schedule B Day -7) and Schedule A Cycle 1/Day 3 or Day 4, Schedule B Cycle 1/Day 8 or 9
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-03814735 80 mg (Schedule A) | PF-03814735 50 mg (Schedule B)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Target Modulation by Phosphohistone H3 (pH3) Expression in Tumor Tissue (IHC)
Description: pH3 expression is a method to enable the quantification of the proliferative potential of tumor cells. Post-dose tumor tissue sampling occurred after FDG-PET. Biopsies were not to be taken from lesions which were used for PET analysis and were to be taken between 1 and 6 hours after study drug administration. Collected in the expanded MTD cohort only (≥ 10 participants in Sch A 80 mg and Sch B 50 mg groups).
Time Frame: Schedule A Cycle 1 or Cycle 2 /Day 4 or Day 5, Schedule B Cycle 1/Day 9 or Day 10
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | PF-03814735 80 mg (Schedule A) | PF-03814735 50 mg (Schedule B)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Objective Tumor Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: Every 2 cycles (each cycle=21 days) until disease progression or participant discontinuation; maximum follow-up was from baseline up to 12 cycles
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Number; unit: participants
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Time to Progression
Description: Time to Progression defined as the time from the date of enrollment to the date progressive disease first reported. If tumor progression data included more than 1 date, the first date was to be used. TTP = (first date of tumor progression - date of enrollment + 1). Progressive disease: ≥20% increase in sum LD of target lesions from smallest sum LD recorded since treatment start or appearance of ≥1 new lesions.
Time Frame: Baseline, every 2 cycles (each cycle=21 days) until disease progression or participant discontinuation; maximum follow-up was from baseline up to 12 cycles
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Number; unit: months
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Duration of Response
Description: Duration of responses based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: as for outcome 12
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Number; unit: months
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Germ Line Polymorphism of Candidate Genes Targeted by PF-03814735
Description: Percentage of germ line polymorphism cell expression in relation to clinical response. Responses include CR: disappearance of all target lesions; PR: ≥30% decrease in sum of LD of target lesions referencing baseline sum LD; Progressive disease: ≥20% increase in sum LD of target lesions from smallest sum LD recorded since Tx start or appearance of ≥1 new lesions; Stable disease: neither sufficient shrinkage to=PR nor sufficient increase to=PD during first 6 weeks after Tx start referencing smallest sum LD since Tx start.
Time Frame: Schedule A Cycle 1 or Cycle 2 /Day 4 or Day 5, Schedule B Cycle 1/Day 9 or Day 10 (each cycle=21 days)
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Number; unit: percentage of cells
Arm/Group | PF-03814735 80 mg (Schedule A) | PF-03814735 50 mg (Schedule B)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Aurora Gene Somatic Mutations/Amplification and Pathway Genes in Tumor Tissue
Description: Percentage of aurora gene somatic mutations/amplification and pathway genes in relation to clinical response. Responses include CR: disappearance of all target lesions; PR: ≥30% decrease in sum of longest dimensions (LD) of target lesions referencing baseline sum LD; Progressive disease: ≥20% increase in sum LD of target lesions from smallest sum LD recorded since Tx start or appearance of ≥1 new lesions; Stable disease: neither sufficient shrinkage to=PR nor sufficient increase to=PD during first 6 weeks after Tx start referencing smallest sum LD since Tx start.
Time Frame: Schedule A Cycle 1 or Cycle 2 /Day 4 or Day 5, Schedule B Cycle 1/Day 9 or Day 10 (each cycle=21 days)
Population: Data was not summarized as the development of the compound was discontinued.
Measure: Number; unit: percentage of cells
Arm/Group | PF-03814735 80 mg (Schedule A) | PF-03814735 50 mg (Schedule B)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent events are reported from the first dose of study treatment up to 28 days after last dose of study treatment.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-03814735 5 mg (Schedule A) | PF-03814735 10 mg (Schedule A) | PF-03814735 20 mg (Schedule A) | PF-03814735 40 mg (Schedule A) | PF-03814735 60 mg (Schedule A) | PF-03814735 80 mg (Schedule A) | PF-03814735 100 mg (Schedule A) | PF-03814735 40 mg (Schedule B) | PF-03814735 50 mg (Schedule B) | PF-03814735 60 mg (Schedule B)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/1 | 1/4 | 1/3 | 4/15 | 2/7 | 0/3 | 5/16 | 0/6
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 4/4 | 3/3 | 15/15 | 7/7 | 3/3 | 15/16 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03814735 5 mg (Schedule A) (N=1) | PF-03814735 10 mg (Schedule A) (N=1) | PF-03814735 20 mg (Schedule A) (N=1) | PF-03814735 40 mg (Schedule A) (N=4) | PF-03814735 60 mg (Schedule A) (N=3) | PF-03814735 80 mg (Schedule A) (N=15) | PF-03814735 100 mg (Schedule A) (N=7) | PF-03814735 40 mg (Schedule B) (N=3) | PF-03814735 50 mg (Schedule B) (N=16) | PF-03814735 60 mg (Schedule B) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03814735 5 mg (Schedule A) (N=1) | PF-03814735 10 mg (Schedule A) (N=1) | PF-03814735 20 mg (Schedule A) (N=1) | PF-03814735 40 mg (Schedule A) (N=4) | PF-03814735 60 mg (Schedule A) (N=3) | PF-03814735 80 mg (Schedule A) (N=15) | PF-03814735 100 mg (Schedule A) (N=7) | PF-03814735 40 mg (Schedule B) (N=3) | PF-03814735 50 mg (Schedule B) (N=16) | PF-03814735 60 mg (Schedule B) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glare (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 6 | 1 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 2 | 7 | 4 | 2 | 7 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 7 | 4 | 1 | 5 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 1 | 5 | 2 | 0 | 4 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 9 | 3 | 1 | 5 | 4
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 6 | 2 | 1 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 0 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.